CLINICAL TRIAL: NCT01375374
Title: Multicenter, Open-label, Single-arm Study to Evaluate Hormone and Lipid Levels in Male Subjects With Partial-onset Seizures After a Switch of Treatment From Carbamazepine as Adjunctive Treatment to Levetiracetam to Lacosamide as Adjunctive Treatment to Levetiracetam
Brief Title: Hormonal and Lipid Levels in Male Subjects After a Switch From Carbamazepine to Lacosamide
Acronym: VICTOR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow progress despite recruitment boosting efforts e.g., expert advice obtained from leading study center Investigators; decision thus made to terminate.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0978; 2010-022534-84 (EudraCT Number)
Record Dates: First submitted 2011-05-09; First posted 2011-06-17 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy, Partial
Keywords: Vimpat; Partial seizures; Carbamazepine; Hormone levels; Lipid levels; Lacosamide
MeSH Terms: conditions — Epilepsies, Partial; Seizures | interventions — Lacosamide; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): commercial 50 mg (pinkish) and 100 mg (yellow) tablets
  Interventions: Drug: Lacosamide; Drug: Levetiracetam

INTERVENTIONS:
Drug: Lacosamide — 4-Week Titration Period: start dose Lacosamide (LCM) is 100 mg/day - up-titration of 100 mg/week LCM 8-Week Maintenance Period: dose can change first 4 weeks with 100 mg/week, must remain between 300 mg/day and 600 mg/day. Dose must remain stable last 4 weeks.
  Other Names: Vimpat
Drug: Levetiracetam — Levetiracetam (LEV) is taken at a stable dose 30 days before study entry and is ≥ 1000 mg/day at the first visit. The LEV dose may not be changed at any time.
  Other Names: Keppra

SUMMARY:
The purpose of the trial is to investigate whether changes in lipids and hormonal parameters can be observed in blood when Carbamazepine treatment is replaced with Lacosamide treatment, while Levetiracetam treatment remains unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Male subject with diagnosis of Epilepsy with Partial-Onset Seizures
* Subject only taking Levetiracetam in combination with Carbamazepine as adjunctive treatment for Epilepsy

Exclusion Criteria:

* Subject is taking another Anti-Epileptic Drug (AED) than Carbamazepine (CBZ) and Levetiracetam (LEV)
* Subject is taking lipid lowering agents
* Subject is taking enzyme inducers

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (7):
- Austria (2):
  - 11, Innsbruck
  - 12, Salzburg
- Germany (3):
  - 2, Bielefeld
  - 1, Bonn
  - 5, Erlangen
- Spain (2):
  - 22, Alcorcón
  - 20, Santiago de Compostela

REFERENCES:
- [Derived] Elger CE, Rademacher M, Brandt C, Elmoufti S, Dedeken P, Eckhardt K, Tennigkeit F, De Backer M. Changes in hormone and lipid levels in male patients with focal seizures when switched from carbamazepine to lacosamide as adjunctive treatment to levetiracetam: A small phase IIIb, prospective, multicenter, open-label trial. Epilepsy Behav. 2016 Sep;62:1-5. doi: 10.1016/j.yebeh.2016.05.023. Epub 2016 Jul 15. PMID 27423106
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites across Austria (1 site), Germany (3 sites), and Spain (1 site).
Pre-assignment Details: The study consisted of a 1-week Screening Period, a 12-week Treatment Period (comprised of a 4-week Titration Period and an 8-week Maintenance Period), and a Taper/Safety Follow-Up Period 3 to 4 weeks in duration.
Groups:
- Lacosamide: commercial 50 mg (pinkish) and 100 mg (yellow) tablets
  * Lacosamide: 4-week Titration Period: start dose Lacosamide (LCM) was 100 mg/day - up-titration of 100 mg/week LCM.
    8-week Maintenance Period: dose could change first 4 weeks with 100 mg/week, needed to remain between 300 mg/day and 600 mg/day. Dose needed to remain stable last 4 weeks.
  * Levetiracetam: Levetiracetam (LEV) was taken at a stable dose 30 days before study entry and was ≥ 1000 mg/day at the first visit. The LEV dose could not be changed at any time.
Period: Overall Study
Arm/Group | Lacosamide
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Safety Set (SS). The SS consists of all patients who received at least 1 dose of Lacosamide.
Arm/Group | Lacosamide
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (5.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Black or African American | 0
  Native Hawaiin or other Pacific Islander | 0
  White | 9
  Other/Mixed | 1
Weight [Mean (Standard Deviation); unit: kilograms] | 82.81 (16.25)
Height [Mean (Standard Deviation); unit: centimeters] | 178.05 (10.14)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] | 25.89 (3.01)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Sex Hormone Binding Globulin (SHBG) From Baseline to Treatment Period End (Comprised of a 4-week Titration Period and an 8-week Maintenance Period)
Description: Due to premature termination of enrollment prior to achieving the planned sample size (a total of 28 subjects), this primary safety variable was assessed for descriptive purposes only. A negative value indicates an improvement.
Time Frame: From Day 1 (Baseline) to Day 84 (Treatment Period End)
Population: The Analysis Population refers to the Safety Set (SS). The SS consists of all subjects who received at least 1 dose of Lacosamide.
Measure: Median (Full Range); unit: nmol/L
Arm/Group | Lacosamide
Number analyzed (Participants) | 10
nmol/L | -12.80 [-20.3 to 4.9]

2. Secondary Outcome: Change in Sex Hormone Calculated Free Androgen Index Levels From Baseline to Treatment Period End (Comprised of a 4-week Titration Period and an 8-week Maintenance Period)
Description: The change in sex hormone calculated free androgen index (100 x Testosterone/sex hormone binding globulin) levels from Baseline to the end of Maintenance Period was summarized descriptively by visit. A negative value indicates an improvement.
Time Frame: From Day 1 (Baseline) to Day 84 (Treatment Period End)
Population: as for outcome 1
Measure: Median (Full Range); unit: Free Androgen Index
Arm/Group | Lacosamide
Number analyzed (Participants) | 10
Free Androgen Index | 9.493 [2.39 to 26.46]

3. Secondary Outcome: Change in Serum Thyroid Hormone Free Thyroxine Level From Baseline to Treatment Period End (Comprised of a 4-week Titration Period and an 8-week Maintenance Period)
Description: The change in the serum thyroid hormone free thyroxine level from Baseline to the end of the Maintenance Period was summarized descriptively by visit.
Time Frame: From Day 1 (Baseline) to Day 84 (Treatment Period End)
Population: as for outcome 1
Measure: Median (Full Range); unit: pmol/L
Arm/Group | Lacosamide
Number analyzed (Participants) | 10
pmol/L | 2.70 [1.5 to 5.5]

4. Secondary Outcome: Change in Total Cholesterol Level From Baseline to Treatment Period End (Comprised of a 4-week Titration Period and an 8-week Maintenance Period)
Description: The change in total cholesterol levels from Baseline to the end of the Maintenance Period was summarized descriptively by visit. A negative value indicates an improvement.
Time Frame: From Day 1 (Baseline) to Day 84 (Treatment Period End)
Population: as for outcome 1
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Lacosamide
Number analyzed (Participants) | 10
mmol/L | -0.540 [-1.46 to 0.11]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Event were reported from Baseline until the Safety Follow-up Visit (two weeks after end of Treatment Period).
Description: Only Treatment Emergent Adverse Events are presented.
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=11)
Fatigue (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The results of this study are limited due to the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days